CLINICAL TRIAL: NCT05969431
Title: Hair Cortisol as Marker of Chronic Stress in Preterm and Term Fathers - Fathair-study
Status: Recruiting | Type: Observational
Sponsor: University of Cologne (Other)
Collaborators: University of Siegen (Unknown)
Responsible Party: Principal Investigator, Katrin Mehler, Associate Professor, University of Cologne
Other Study IDs: 23-114058
Record Dates: First submitted 2023-07-24; First posted 2023-08-01 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Stress, Psychological; Father-Child Relations; Premature Birth
MeSH Terms: conditions — Stress, Psychological; Premature Birth | interventions — Pain Measurement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — A hair sample will be taken from the back of the father's head (a thin strand of hair, approximately a total diameter of 3-5 mm). From this sample only the cortisol level will be measured.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- fathers of mature infants: Fathers of newborns' above 37 weeks of gestation
  Interventions: Diagnostic Test: measurement of cortisol level
- fathers of moderate and late preterm infants: Fathers of moderate and late preterm infants, i.e. gestational age from 32 0/7 to 36 6/7 weeks of gestation.
  Interventions: Diagnostic Test: measurement of cortisol level
- fathers of very low birth weight preterm infants: Fathers of very low birth weight preterm infants, i.e. gestational age from 22 0/7 to 31 6/7 weeks of gestation and with a birth weight below 1500 g.
  Interventions: Diagnostic Test: measurement of cortisol level

INTERVENTIONS:
Diagnostic Test: measurement of cortisol level — We will measure the cortisol level from the hair sample of the father at three time points. Furthermore the father will answer questionnaires at three time points and the paternal sensitivity is measured once.
  Other Names: questionnaire

SUMMARY:
The goal of this observational study is to compare the paternal hair cortisol as a marker for chronic stress in prematurely born children to maturely born children.

The main questions it aims to answer are:

* How differ the cortisol level between groups?
* How change the cortisol level over time?
* Are there secondary outcomes associated to the cortisol level of fathers? Participants will give a hair sample to analyse the cortisol level and fill out questionnaires at three time points. At six months of the infant's age, the investigators will also measure the paternal sensitivity.

DETAILED DESCRIPTION:
For expectant parents, the birth of a child is often a stressful situation. In the case of a premature birth, the psychological stress is usually increased because the parents frequently could not prepare for the birth. Therefore, the researcher would like to investigate this stress of fathers of newborn children.

For this purpose, the stress hormone cortisol in the fathers' hair will be analysed and questionnaires on the fathers' mental health will be collected. Subsequently, the differences between fathers of prematurely born and of maturely born children will be compared.

The investigators will do the analyses at three time points: the first time point will be at the first week after birth, the second three months and the third six months after birth. At six months of the infant's age, additionally the paternal sensitivity will be measured.

The compared groups will differ with respect to gestational age: Group 1 includes preterm infants with a gestational age below 32 weeks and a birth weight <1500 grams (very low birthweight infants), group 2 preterm infants with a gestational age between 32 0/7 to 36 6/7 (moderate and late preterm infants) and group 3 consists of mature infants (over 37 weeks gestational age).

ELIGIBILITY:
Inclusion Criteria:

* Premature or mature infant (22 0/7 to 42 0/7 weeks of gestation)
* For mature infants (37 0/7 to 42 0/7 weeks of gestation) undisturbed neonatal period
* No severe malformations or genetic diseases of the newborn child
* Sufficient knowledge of German of the father
* written consent of the custodial parents

Exclusion Criteria:

* adoptive or foster paternity
* hair length below 3 cm at the posterior vertex region of the back of the father's head
* endocrine disorders, especially of the adrenocortical system (e.g. Cushing syndrome, adrenal insufficiency)
* taking steroidal medications or other drugs that affect the activity of the hypothalamic-pituitary-adrenocortical system
* paternal psychological or severe physical illness

Ages: 1 Day to 7 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Fathers of newborns born at the university hospital of Cologne
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
hair cortisol level | first week after birth, 3 and 6 months after birth
  The level of cortisol will be measured in the hair of the fathers by liquid chromatography with tandem mass spectrometry. This test is validated in human hair and the current gold standard method in hair steroid analysis. The analytic procedure follows a published laboratory protocol that has excellent sensitivity, specificity and reliability.

SECONDARY OUTCOMES:
Cortisone, testosterone, progesterone, dehydroepiandrosterone level in the paternal hair | first week after birth, 3 and 6 months after birth
  The level of these hormones (cortisone, testosterone, progesterone, dehydroepiandrosterone) will be measured in the hair of the fathers by liquid chromatography with tandem mass spectrometry. This test is validated in human hair and the current gold standard method in hair hormone analysis. The analytic procedure follows a published laboratory protocol that has excellent sensitivity, specificity and reliability.
paternal sensitivity | 6 months after birth
  The paternal sensitivity and the father-child-interaction will be measured during a five-minute-videotape of the father changing the infants' diapers and playing with the infant. The paternal sensitivity will be measured by a 9-point scale. The score can range from 1 to 9, where 1 means lack of sensitivity and 9 means very sensitive. The classification is a validated tool and is done by two trained and reliable evaluators from the Department of Developmental Science and Special Education. The evaluators are blinded.
father-child-interaction | six months of age
  The father-infant-interaction is investigated during the same video as the paternal sensitivity using Mannheim Rating Scales by a blinded psychologist. Mannheim Rating Scale is a good validated standardized observation instrument. Stimulation and response from the father as well from the infant are being recorded. Different communication channels can be used by father and child (vocal, facial or motor). All behaviors are analyzed at intervals of five seconds (event coding). The values are formed from the sum of the coded events. The scale ranges from 0 to 60. If there is no interaction, the scale is 0. If there is an interaction in each interval (every 5 seconds in a 5 minute videotape), the scale is 60. The father-child interaction is better if the scale is higher.
paternal depression | first week, 3 and 6 months after birth
  Paternal depression is assessed with the Edinburgh Postnatal Depression Scale (EPDS). It is a self-report questionnaire to measure depressive symptoms especially after birth and it consists of 10 questions. For each question the response choice are assigned point values (how often a symptom occurred during the last week). The point values are summed to a total measure score. The score ranges from 0 to 30. Zero points represents no symptoms of depression, a score of 13 or higher is interpreted to indicate a risk of depression.
socioeconomic status | first week after birth
  There will be questions to the household income per month, the parents' highest school-leaving certificate and the housing situation
social support | three months after birth
  Social support is assessed with the short German version of the questionnaire on social support (F-SozU K-22). The questionnaire records the subjectively perceived or anticipated support from the social environment. There are 22 items and the test person can indicate the degree of agreement on a five-level Likert scale (from 1 = does not apply to 5 = applies completely). The scale ranges from a minimum of 22 points to a maximum of 110 points. The higher the score, the better the subjectively perceived or anticipated support.
impact of event scale | six months after birth
  Symptoms for post-traumatic stress is assessed with the impact of event scale - revised (IES-R). It is a self-report questionnaire and consists of 22 questions. For each question the response choice are assigned point values (how often a symptom occurred during the last week). The sub-scale values are summed by the corresponding sub-scale items. The three sub-scales are: intrusion, avoidance and hyperarousal. The overall result is calculated by a formula. The score ranges from -4,36 to 2,99. A result above 0 is interpreted to indicate a risk for post-traumatic stress disorder.
Parental Bonding | first week, 3 and 6 months after birth
  Parental Bonding is assessed with the parental bonding questionnaire (PBQ). It consists of 25 items and each item is rated on a scale from 0 to 3 points (response range from "very like" to "very unlike"). There are four sub-scales and the point values of each sub-scale are summed to a total measure score. The four sub-scales are: impaired bonding, rejection and anger, anxiety about care, risk of abuse. The higher the score, the higher the risk of a disorder in each area of the sub-scale.
Parental Stress | six months after birth
  Parental stress is assessed with the German form of the parenting stress index (PSI).
  It consists of 48 items. The test person can indicate the degree of agreement on a five-level Likert scale (from 1 = does not apply to 5 = applies completely). There are 12 subscales, each consisting of 4 items and the points on the Likert scale are added. In each subscale there can be a minimum of 4 and a maximum of 20 points. The higher the score, the higher the parental stress.
Parental Stress | first week, 3 and 6 months after birth
  The perceived parental stress is assessed by the German version from the perceived stress scale (PSS-10). It is a self-report questionnaire to measure symptoms of stress and it consists of 10 questions. For each question the response choice are assigned point values (how often a symptom occurred during the last month). There are two subscales (perceived helplessness and perceived self-efficacy). The subscale perceived self-efficacy are reversed score for the total score. The point values of both subscales are summed to a total measure score. The score ranges from 0 to 50. Zero points represents no symptoms of stress, higher scores reflect greater levels of stress.

CONTACTS AND LOCATIONS:
Overall Officials: Katrin Mehler, PD Dr., Principal Investigator — University of Cologne
Locations (1):
- University Hospital of Cologne, Cologne, Northrhine-westfalia, Germany

IPD SHARING:
Plan to Share IPD: No